CLINICAL TRIAL: NCT00465790
Title: GENomic Biomarkers for PARKinson's Disease
Brief Title: Research of Biomarkers in Parkinson Disease
Acronym: Genepark
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: C06-56; 2007-A00208-45
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Progressive Supranuclear Palsy; Huntington Disease; Dystonia; Diffuse Lewy Body Disease
Keywords: biomarkers; neuroimaging; genetics; PET; Genetic and Idiopathic Parkinson; Multiple Systemic Atrophy; Huntington; Dopa Responsive Dystonia
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive; Huntington Disease; Dystonia; Lewy Body Disease; Dystonia, Dopa-responsive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The main goal of the GENEPARK consortium is to employ innovative haemogenomic approaches to determine gene expression profiles specific for genetic and idiopathic Parkinson's disease (PD) patients. These gene expression signatures will be utilised clinically as non-invasive diagnostic tests for PD. The sensitivity of the newly developed diagnostic test will be determined by extensive validations on an independent cohort of PD patients, whereas the specificity will be assessed by testing patients with atypical parkinsonisms, including multiple system atrophy, progressive supranuclear palsy and diffuse Lewy body disease. In order to test the specificity of the diagnostic set in other disorders that affect basal ganglia, Huntington's disease and dopa responsive dystonia patients will be analysed. The second objective of the proposal is to determine correlations between gene expression signatures and different stages of PD and thus provide the basis for early diagnosis and monitoring of disease progression. These changes in blood gene expression will be correlated with alterations detected by neuroimaging in the brain of PD patients. Such combinations of molecular and morphological markers of disease may ultimately facilitate the selection and monitoring of neuroprotective therapies for PD. Finally, GENEPARK aims to develop new bioinformatic software tools for selection of genomic biomarkers using microarray data. A set of established computational tools will be applied and novel methods, some of them based on mechanistic modelling of the neurodegenerative diseases, will be developed in order to study the advantages and limitations of the different methodologies.

With special emphasis on the careful clinical selection of patients and sufficient power regarding patient numbers, as well as extensive quality control and validation of the data, GENEPARK aims to develop a standardised approach to development and validation of haemogenomic biomarkers of disease.

DETAILED DESCRIPTION:
Employ innovative haemogenomic approaches to determine gene expression signatures specific for idiopathic Parkinson's disease (PD). There is currently no specific clinical or laboratory diagnostic test available for PD. In GENEPARK, blood samples from patients with genetic PD and idiopathic PD will be analysed by microarrays to identify gene expression signatures specific for PD. The specificity of the new biomarkers for PD will be tested by the analysis of patients with atypical parkinsonisms, including multiple system atrophy (MSA), progressive supranuclear palsy (PSP) and diffuse Lewy body disease (DLBD), as well as in patients with other basal ganglia disorders such as Huntington's disease (HD) and dopa responsive dystonia (DRD). The validated gene expression signatures will be utilised to develop a new test for diagnosis of idiopathic PD. Determine correlation between gene expression signatures and different stages of PD.

Gene expression in presymptomatic and symptomatic patients with genetic forms of PD as well as patients in various stages of idiopathic PD will be analysed to identify gene expression signatures specific for various stages of the disease. It should be emphasised that since no clinical measures are present in presymptomatic genetic PD such molecular markers could serve as surrogate markers to monitor therapeutic efficacy of possible preventive treatments in PD. Determine correlations between gene expression signatures and morphological evidence of neurodegenerative process in PD brain as determined by neuroimaging. Gene expression signatures identified in blood samples will be correlated with changes in brain as detected by neuroimaging in PD patients. Such correlations of molecular and morphological markers of disease will facilitate the selection of blood markers in relation to disease progression. Moreover, molecular and morphological markers of disease progression could be utilised in combination for monitoring the effects of new neuroprotective therapies for PD. Develop standardised approaches to development and validation of haemogenomic biomarkers.

This objective will be achieved by the special emphasis on careful clinical selection of patients, sufficient power regarding patient numbers, as well as extensive quality control and validation of the data. Develop new bioinformatic software tools for selection of genomic biomarkers using microarray data. The aim of the GENEPARK is to develop the theoretical foundations and to build the software tools for sample classification and selection of genomic biomarkers using microarray data. The established computational tools and novel methods developed within the GENEPARK will be applied to the patient data to study advantages and limitations of different methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Ability to understand the aim of the study
* Ability to sign the consent form

Exclusion Criteria:

* Non ability to understand the aim of the study
* Non ability to sign the consent form
* To be over 18

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease and related
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2007-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Borut Perterlin, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (5):
- Meditterranean Institute for Life Sciences, Split, Croatia
- INSERM Unit 679, Paris, France
- Germany (2):
  - University of Lübeck and Neuroimage Nord, Lübeck
  - University Hospital Tübingen, Tübingen
- University Medical Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- See also: Related Info — http://www.inserm.fr